CLINICAL TRIAL: NCT04192240
Title: Immediate Effects of Lower Limb Loading Training During Sit-to-stand and Stepping With and Without External Feedback in Ambulatory Individuals With Stroke
Brief Title: Weight-bearing Training in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr., Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MSD60I0015
Record Dates: First submitted 2019-03-10; First posted 2019-12-10 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: cerebrovascular disease; rehabilitation; walking; balance; mobility
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WB Training with external feedback (Experimental): WB during sit-to-stand with external feedback for 10 minute and then, WB during stepping training with external feedback for 10 minutes. After training, subjects will walk overground for 10 minutes.
  Interventions: Other: WB Training with external feedback
- WB Training without external feedback (Active Comparator): WB during sit-to-stand without external feedback for 10 minute and then, WB during stepping training without external feedback for 10 minutes. After training, subjects will walk overground for 10 minutes.
  Interventions: Other: WB Training without external feedback

INTERVENTIONS:
Other: WB Training with external feedback — WB during sit-to-stand and stepping with external feedback, follow by overground walking.
  Arms: WB Training with external feedback
Other: WB Training without external feedback — WB during sit-to-stand and stepping without external feedback, follow by overground walking.
  Arms: WB Training without external feedback

SUMMARY:
1. Are there differences in weight-bearing (WB) and WB symmetry immediately following STS and stepping training with or without using external feedback in ambulatory patients with stroke?

1. Are there differences in mobility immediately following STS and stepping training with or without using external feedback in ambulatory patients with stroke?

DETAILED DESCRIPTION:
Subjects are patients with stroke, the age of over 40 years to 74 years, both males and females who are able to walk independently at least 10 meters. Most of them will be recruited from a tertiary rehabilitation center and communities. Subjects have to participate in STS and stepping training with and without using the external feedback for 1 time/condition with a wash-out period for 2 weeks (crossover design). The outcomes will be measured in terms of WB ability during STS and stepping, walking speed, and balance ability.

The primary outcomes were WB ability on the affected limb and WB symmetry. Secondary outcomes were walking speed and balance ability.

ELIGIBILITY:
Inclusion Criteria:

* Independent ambulatory patients with chronic stroke (post-stroke time more than 6 months)
* Age at least 40 years to 74 years
* Body mass index (BMI) between 18.5- 29.9 kg/m^2
* Ability of independent walking over at least 10 meters with or without a walking device
* Ability to rise from a chair with or without using their arms
* Ability to follow a command used in the study

Exclusion Criteria:

any conditions that may affect ambulatory ability or ability to participate in the study, such as

* Auditory or visual deficits that are unable to be corrected by a hearing aid, glasses or contact lens
* Musculoskeletal pain with a pain scale more than 5 out of 10 on a visual analog scale (VAS)
* Deformity in the limbs or spine that affect ambulatory ability
* Modified Ashworth Scale (MAS) more 2 score
* Unstable cardiovascular, orthopedics, musculoskeletal, or neurological disease other than stroke.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Weight-bearing (WB) ability and WB symmetry | Prior to and immediately after complete training program in one session

SECONDARY OUTCOMES:
Walking speed using the 10 meter-walk test (10MWT) | Prior to and immediately after complete training program in one session
Dynamic balance control using the Timed up and go test (TUGT) | Prior to and immediately after complete training program in one session

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, Principal Investigator — School of physical therapy, Faculty of Associated medical sciences, Khon Kaen University
Locations (1):
- Faculty of Associated Medical Science, Nai Muang, KhonKaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Boukadida A, Piotte F, Dehail P, Nadeau S. Determinants of sit-to-stand tasks in individuals with hemiparesis post stroke: A review. Ann Phys Rehabil Med. 2015 Jun;58(3):167-72. doi: 10.1016/j.rehab.2015.04.007. Epub 2015 May 23. PMID 26004813
- [Result] Lomaglio MJ, Eng JJ. Muscle strength and weight-bearing symmetry relate to sit-to-stand performance in individuals with stroke. Gait Posture. 2005 Oct;22(2):126-31. doi: 10.1016/j.gaitpost.2004.08.002. PMID 16139747
- [Result] Park GD, Choi JU, Kim YM. The effects of multidirectional stepping training on balance, gait ability, and falls efficacy following stroke. J Phys Ther Sci. 2016 Jan;28(1):82-6. doi: 10.1589/jpts.28.82. Epub 2016 Jan 30. PMID 26957733
- [Result] Tsaklis PV, Grooten WJ, Franzen E. Effects of weight-shift training on balance control and weight distribution in chronic stroke: a pilot study. Top Stroke Rehabil. 2012 Jan-Feb;19(1):23-31. doi: 10.1310/tsr1901-23. PMID 22306625